CLINICAL TRIAL: NCT04678076
Title: A Bioequivalence Study of a Test Formulation of Ketoprofen Oral Gel 25 mg Versus a Marketed Reference of Ketoprofen Lysine Salt as Granules for Oral Solution (80 mg Bipartite Sachet, Half Sachet) After Single Dose Administration Under Fed Conditions to Healthy Male and Female Subjects
Brief Title: Bioequivalence of Ketoprofen Oral Gel vs Ketoprofen Lysine Salt as Granules for Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 145(B)WO17389; CRO-PK-18-326 (Other: CROSS Research)
Record Dates: First submitted 2020-12-09; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: ketoprofen; oral gel; ketoprofen Lysine Salt as granules; bioequivalence
MeSH Terms: interventions — ketoprofen lysine

STUDY DESIGN:
Intervention Model Description: Single dose, open-label, randomised, two-period, two-way cross-over, two-stage bioequivalence study.
Masking Description: No masking procedure will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketoprofen 25mg/5ml oral gel stick pack (Experimental): Single dose of ketoprofen 25mg/5ml oral gel stick pack will be administered to healthy volunteers under fed conditions in two consecutive study periods with a wash-out interval of at least 7 days between the two administrations.
  Interventions: Drug: Ketoprofen Lysine
- OKi 80 mg granules for oral solution (bipartite sachet) (Active Comparator): Single dose of half sachet containing 40 mg of ketoprofen lysine salt (corresponding to 25 mg as ketoprofen) will be administered to healthy volunteers under fed conditions in two consecutive study periods with a wash-out interval of at least 7 days between the two administrations.
  Interventions: Drug: Ketoprofen Oral Product

INTERVENTIONS:
Drug: Ketoprofen Lysine — A single oral dose of test product - ketoprofen 25 mg/5 ml oral gel stick pack - will be administered to healthy male and female volunteers under fed conditions in two consecutive study periods with a wash-out interval of at least 7 days between the two administrations.
  Arms: ketoprofen 25mg/5ml oral gel stick pack
Drug: Ketoprofen Oral Product — A single oral dose of reference product as a single dose of half of a bipartite sachet of OKi® 80 mg granules for oral solution will be administered to healthy male and female volunteers under fed conditions in two consecutive study periods with a wash-out interval of at least 7 days between the two administrations.
  Other Names: OKI 80 mg
  Arms: OKi 80 mg granules for oral solution (bipartite sachet)

SUMMARY:
This is a single dose, open-label, randomised, two period, two-way cross-over, two stage bioequivalenve study with the aim to investigate the bioequivalence between a new formulation of ketoprofen 25 mg versus OKI 80 mg granules for oral solution (half sachet), after single dose administration in two consecutive periods to healthy voluteers under fed conditions.

DETAILED DESCRIPTION:
The present bioequivalence phase I study has been designed to compare the bioavailability and the concentration-time profile of the new immediate release oral gel formulation of ketoprofen 25 mg with a marketed reference of ketoprofen lysine salt (KLS) as granules for oral solution (80 mg bipartite sachet, half sachet containing 40 mg of KLS, corresponding to 25 mg as ketoprofen), when administered in fed conditions to healthy male and female subjects. The study has been designed under fed conditions since the leaflet of the reference.

A two-stage design has been selected for the present study considering the margin of uncertainty existing over the sample size estimate in order to accomplish the primary study objectives in terms of ketoprofen rate (Cmax) and extent (AUC0-t) of absorption of the two formulations.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: signed written informed consent before inclusion in the study.
* Sex and Age: males/females, 18-55 years old inclusive.
* Body Mass Index (BMI): 18.5-30 kg/m2 inclusive.
* Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg and heart rate 50-90 bpm, measured after 5 min of rest in the sitting position.
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
* Contraception and fertility (females only): females of child-bearing potential and with an active sexual life must be using at least one of the following reliable methods of contraception:

  1. Hormonal oral, implantable, intrauterine device [IUD], transdermal or injectable contraceptives for at least 2 months before the screening visit
  2. A non-hormonal IUD or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
  3. A male sexual partner who agrees to use a male condom with spermicide
  4. A sterile sexual partner
* Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, pregnancy test result must be negative at screening and day -1 of each study period.

Exclusion Criteria:

* Electrocardiogram (ECG 12-leads, supine position): clinically significant abnormalities.
* Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study.
* Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness.
* Allergy: ascertained or presumptive hypersensitivity to the active principles (ketoprofen) and/or formulations' ingredients; history of hypersensitivity to drugs (in particular to NSAIDs) or allergic reactions in general, which the Investigator considers may affect the outcome of the study.
* Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory (including asthma), skin, haematological, endocrine or neurological and autoimmune diseases that may interfere with the aim of the study.
* Medications: medications, including over the counter (OTC) drugs [in particular ketoprofen, acetylsalicylic acid (ASA) and NSAIDs in general], herbal remedies and food supplements for 2 weeks before the start of the study. Paracetamol will be allowed as therapeutic counter-measure for adverse events (AEs) according to the Investigator's opinion. Hormonal contraceptives and hormone replacement therapies for females will be allowed.
* Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study (date of the informed consent signature).
* Blood donation: blood donations for 3 months before this study.
* Drug, alcohol, caffeine, tobacco: history of drug, alcohol [> 1 drink/day for females and > 2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015-2020, caffeine (more of 5 cups coffee/tea/day) or tobacco abuse (more or equal of 6 cigarettes/day).
* Drug test: positive result at the drug test at screening or day -1 of each study period.
* Alcohol test: positive alcohol breath test at day -1 of each study period.
* Diet: abnormal diets (< 1600 or > 3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians.
* Pregnancy (females only): positive or missing pregnancy test at screening or day -1 of each study period; pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of ketoprofen | pre-dose (0), 20, 40 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  to evaluate the rate (Cmax) of absorption of ketoprofen after single oral dose of test and reference.
Area under the concentration-time curve 0-t | pre-dose (0), 20, 40 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  to evaluate the extent (AUC0-t) of absorption after single oral dose of test and reference

SECONDARY OUTCOMES:
Time to achieve Cmax | pre-dose (0), 20, 40 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  to evaluate Tmax after single oral dose of test and reference products
t1/2 | pre-dose (0), 20, 40 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  to evaluate Half-life after single oral dose of test and reference products
tlag after single oral dose of test and reference products | pre-dose (0), 20, 40 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  to evaluate Lag-time observed from the dosing time point prior to that of the first measurable plasma concentration
AUC0-∞ and residual area of ketoprofen derived from plasma concentrations after single oral dose of test and reference products; | pre-dose (0), 20, 40 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Area under the concentration-time curve extrapolated to infinity
Treatment-Emergent Adverse Events | through study completion, an average two weeks
  to evaluate number of TEAEs and percentage of subjects with TEAEs
Blood pressure measurement | pre-dose, 45 minutes and 24 hours post dose
  to assess diastolic and systolic blood pressure after 5 min of rest (sitting position).
Heart rate | pre-dose, 45 minutes and 24 hours post dose
  to assess heart rate after 5 min of rest (sitting position).

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research S.A., Phase I Unit, Via F.A. Giorgioli 14 CH-6864 Arzo, Switzerland
Locations (1):
- CROSS Research S.A., Phase I Unit,, Arzo, Switzerland